CLINICAL TRIAL: NCT00001963
Title: Vascular Effects of Endothelium-Derived Versus Hemoglobin-Transported Nitric Oxide in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000031; 00-H-0031
Record Dates: First submitted 2000-01-18; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Diabetes Mellitus; Healthy; Hypercholesterolemia; Hypertension
Keywords: Blood Flow; Exercise; Microcirculation; S-nitrosohemoglobin; Vasodilation; Healthy Volunteer
MeSH Terms: conditions — Diabetes Mellitus; Hypercholesterolemia; Hypertension; Motor Activity; Aneurysm

INTERVENTIONS:
Procedure: hemoglobin-transported nitric oxide

SUMMARY:
Nitric oxide (NO) is a soluble gas, continuously synthesized by the endothelium, that contributes importantly to vasodilator tone of the coronary and systemic circulations by activating guanylyl cyclase in vascular smooth muscle, causing relaxation. Although regional synthesis of NO by the endothelium contributes to local vasodilator tone, Stamler and co-workers have proposed that regional vascular tone may also be regulated by NO transported from the lungs by hemoglobin as a consequence of enhanced binding of NO to reactive thiols of oxygenated hemoglobin. This study is designed to determine the contribution of hemoglobin-transported NO to forearm microvascular dilator tone in healthy subjects at rest and during regional hypoxia associated with forearm exercise stress, with measurements made before and after regional blockade of endothelial NO synthesis. Findings in this study may be relevant to understanding the physiological contribution and therapeutic potential of hemoglobin-transported NO in the regulation of vasodilator tone in diseases and conditions associated with regional endothelial dysfunction and reduced endothelial NO bioactivity (e.g., hypertension, diabetes mellitus, hypercholesterolemia, cigarette smoking, and estrogen deficiency).

DETAILED DESCRIPTION:
Nitric oxide (NO) is a soluble gas, continuously synthesized by the endothelium, that contributes importantly to vasodilator tone of the coronary and systemic circulations by activating guanylyl cyclase in vascular smooth muscle, causing relaxation. Although regional synthesis of NO by the endothelium contributes to local vasodilator tone, Stamler and co-workers have proposed that regional vascular tone may also be regulated by NO transported from the lungs by hemoglobin as a consequence of enhanced binding of NO to reactive thiols of oxygenated hemoglobin. This study is designed to determine the contribution of hemoglobin-transported NO to forearm microvascular dilator tone in healthy subjects at rest and during regional hypoxia associated with forearm exercise stress, with measurements made before and after regional blockade of endothelial NO synthesis. Findings in this study may be relevant to understanding the physiological contribution and therapeutic potential of hemoglobin-transported NO in the regulation of vasodilator tone in diseases and conditions associated with regional endothelial dysfunction and reduced endothelial NO bioactivity (e.g., hypertension, diabetes mellitus, hypercholesterolemia, cigarette smoking, and estrogen deficiency).

ELIGIBILITY:
All volunteer subjects must be between 21 and 75 years of age, in good health, and must have provided informed, written consent for participation in this study.

No subjects with a history or evidence of present or past hypertension (blood pressure greater than 145/95 mmHg), hypercholesterolemia (LDL cholesterol greater than 130 mg/dL), diabetes mellitus (fasting blood glucose greater than 120 mg/dL), smoking within 2 years, cardiac disease, peripheral vascular disease, coagulopathy, or any other disease predisposing to vasculitis or Raynaud's phenomenon.

No volunteer subject will be allowed to take any medication (oral contraceptive agents are allowed) or vitamin supplements for at least one month prior to study and will not be allowed to take aspirin for one week prior to study.

Pregnancy testing will be required of all women of reproductive age to exclude current pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28
Dates: Start 1999-12; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jia L, Bonaventura C, Bonaventura J, Stamler JS. S-nitrosohaemoglobin: a dynamic activity of blood involved in vascular control. Nature. 1996 Mar 21;380(6571):221-6. doi: 10.1038/380221a0. PMID 8637569
- [Background] Gow AJ, Stamler JS. Reactions between nitric oxide and haemoglobin under physiological conditions. Nature. 1998 Jan 8;391(6663):169-73. doi: 10.1038/34402. PMID 9428761
- [Background] Palmer RM, Ashton DS, Moncada S. Vascular endothelial cells synthesize nitric oxide from L-arginine. Nature. 1988 Jun 16;333(6174):664-6. doi: 10.1038/333664a0. PMID 3131684